CLINICAL TRIAL: NCT06377800
Title: Effects Of Navicular Mobilization In Patients With Planter Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01801 Kainat Fatima
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Plantar Fascitis
Keywords: Planter Fasciitis; Foot Navicular bone; Mobilization,; Flat Foot
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- navicular mobilization along with conventional therapy. (Experimental): In the prone position, when the foot is stabilized by a towel underneath, navicular mobilization is administered. The therapist's fixing hand wraps the calcaneus, grasps the talus bone, and fixes it.
  By placing the thumb on the plantar surface of the foot and pushing with the thumb of the other hand in a dorsal direction, navicular mobilization is provided.
  This dorsal glide will be given with 2 sets of 5 minutes. Each session will be of 30 minutes.
  Interventions: Other: navicular mobilization along conventional therapy.
- conventional therapy (Other): ultrasound therapy at 1.5 w/cm2 for 7 minutes in continuous mode at a 3MHz frequency. Stretching targets the medial arch and surrounding muscles like calf and tibialis posterior with exercises such as arch lift, heel raise, towel pickup, and toe lift. Additionally, strengthening exercises for intrinsic foot muscles like standing toe curls and towel toe curls are included. Ice pack application for 10 minutes follows
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: navicular mobilization along conventional therapy. — In the prone position, when the foot is stabilized by a towel underneath, navicular mobilization is administered. The therapist's fixing hand wraps the calcaneus, grasps the talus bone, and fixes it.
  By placing the thumb on the plantar surface of the foot and pushing with the thumb of the other hand in a dorsal direction, navicular mobilization is provided.
  This dorsal glide will be given with 2 sets of 5 minutes. Each session will be of 30 minutes.
  Arms: navicular mobilization along with conventional therapy.
Other: conventional therapy — ultrasound therapy at 1.5 w/cm2 for 7 minutes in continuous mode at a 3MHz frequency. Stretching targets the medial arch and surrounding muscles like calf and tibialis posterior with exercises such as arch lift, heel raise, towel pickup, and toe lift. Additionally, strengthening exercises for intrinsic foot muscles like standing toe curls and towel toe curls are included. Ice pack application for 10 minutes follows
  Arms: conventional therapy

SUMMARY:
The significance of studying the effects of navicular mobilization in patients suffering from plantar fasciitis lies in its potential to provide valuable insights into non-invasive treatment approaches for a common and debilitating foot condition such as flat foot. Understanding how this therapy impacts navicular height, pain and disability of the foot can lead to improved clinical outcomes and a better understanding of the biomechanical factors contributing to plantar fasciitis. Ultimately, this research may help refine treatment strategies and enhance the quality of life for individuals suffering from this condition

DETAILED DESCRIPTION:
The foot is a complex structure comprising numerous bones, muscles, and ligaments that work together to provide support and facilitate movement. It is supported by three arches: the medial longitudinal arch, the lateral longitudinal arch, and the transverse arch. The medial longitudinal arch plays a crucial role in absorbing weight, but issues like ligament laxity and muscle weakness can cause it to shorten, leading to conditions like plantar fasciitis. Plantar fasciitis, a common overuse injury, occurs when the plantar fascia, a fibrous tissue that supports the arch of the foot, becomes inflamed due to repetitive strain, especially during activities that increase its stretch, such as barefoot walking or stair climbing. People with flat feet are more susceptible to plantar fasciitis due to the overstretching of the plantar fascia caused by the lack of arch support.

Navicular drop, a measure of the navicular bone height, also plays a significant role in foot biomechanics and the development of plantar fasciitis. High navicular height leads to increased foot pronation and tension on the plantar fascia, while low navicular height causes overpronation and arch collapse, both of which can result in inflammation of the plantar fascia. Physiotherapists use techniques like navicular mobilization to address issues related to the navicular bone and improve blood circulation, healing, and pain relief in cases of plantar fasciitis. By understanding the biomechanics of the foot and employing targeted interventions, healthcare professionals can help manage and prevent conditions like plantar fasciitis, allowing individuals to maintain optimal foot health and functionality.

ELIGIBILITY:
Inclusion Criteria:

* Plantar fasciitis with flat foot.
* Positive Flat foot cases diagnosed with foot print measurement.
* Unilateral or bilateral involvement with chronic plantar fasciitis
* Diagnosed case of plantar fasciitis will be taken with navicular drop.
* Navicular Drop (ND) of > 10mm

Exclusion Criteria:

* Patients with Peripheral vascular diseases.
* Patients with History of fractures in the lower limb
* Patients with Skin infections and wounds on the foot
* Patients with any neurological deficit involving foot.
* Patients with a history of foot or ankle surgery.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | four weeks
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). According to researches NPRS shows excellent reliability (0.97 and 0.99, respectively) for the measurement of musculoskeletal pain
(Foot Function Index) | four weeks
  Foot function index is a questionnaire used to assess pathological impact on foot with respect to disability, limitations of activity and pain. It consists of 23 questions which are sub divided into three sub scales. These three sub scales are pain, activity limitation and disability.(19) It's scoring is done by adding these scales which range is from 0 to 100. Minimum score is 0 and maximum is 100. Where 0 shows no pain and 100 shows worst pain.
Navicular drop test | four weeks
  Navicular drop test is used to measure static foot assessment in Sagittal plane of navicular tuberosity in neutral state. The tuberosity of the navicular bone is measured in neutral position, relaxed and stance position. Supinated foot showed less than 5mm, neutral foot shows range from 6 to 8mm or 5 to 9mm and pronated foot shows reading from greater than 10 to 15 or greater than 9mm.
Foot print analysis | four weeks
  In this technique, participants created footprints on paper while standing, submerged clean feet a normal foot, while SPI > 1.15 denotes a flat foot. (22) The correlation test and intraclass correlation coefficient showed that I was a valid and reliable in diagnosing flatfoot (0.427, 0.446).

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No